CLINICAL TRIAL: NCT00444353
Title: A Randomized Study of the Safety and Effectiveness of DL6049 (Injectable Poly-l-lactic Acid) Versus Cosmoplast Collagen Implant in the Treatment of Nasolabial Fold Wrinkles (Long Term Follow-up)
Brief Title: DL6049 Versus Cosmoplast in the Treatment of Nasolabial Fold Wrinkles, Long Term Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DL6049-0301LT
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Nasolabial Fold Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: DL6049 (injectable poly-L-lactic acid)

SUMMARY:
This study is being undertaken to:

* evaluate the degree of correction attainable with DL6049 (injectable poly-L-lactic acid)compared to a commercially available CosmoPlast™ Collagen Implant in the treatment of dermal nasolabial fold wrinkles at 13 months following the last application of study treatment.
* Document the types and incidence of adverse events reported with DL6049 (injectable poly-L-lactic acid)compared with CosmoPlast™ Collagen Implant. Long term adverse events will be assessed for an additional 12 months following discharge from the main study in subjects treated with DL6049.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign a statement of IC and HIPAA authorization. In addition subjects must provide a separate release for use of their photographs in publications; any subject has a right to refuse the photo release without jeopardizing their ability to participate in the study.
* Subjects must be 18-75 yrs of age, of any race or sex
* Female subjects must be post-menopausal for at least 1 yr or have had a hysterectomy; or have a had a tubal ligation; or if of child-bearing potential, must agree to use an approved method of birth control throughout the study (i.e, oral/systemic contraceptives, IUD, or spermicide in combination with barrier method of contraception).
* Subjects seeking augmentation therapy for bilateral correction of nasolabial folds. Subjects must have a score of greater than or equal to 2 and less than or equal to 4 on the photo-numeric wrinkle assessment scale (assessed by a blinded evaluator) of both the left and right nasolabial fold at Visit 1.

Exclusion Criteria:

* Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to local anesthetics (e.g.,lidocaine, etc.), bovine collagen, latex, silicone, carmellose, or mannitol.
* Subjects with a known history of keloids or bleeding disorders.
* Subjects with an active inflammatory process in the area to be treated (skin eruptions such as cysts, pimples, rashes, cancerous/pre-cancerous lesions, or any other active skin disease).
* Subjects with active hepatitis within the past year.
* Subjects who are pregnant (confirmation by pregnancy testing),or plan to become pregnant within the study timeframe, or who are nursing.
* Subjects who plan to undergo major facial surgery (e.g., rhinoplasty with or without implant, facelift, congenital defect repair, etc. during the course of the study.
* Subjects with clinically important disease as judged by the investigator within 3 months of the study (e.g., significant lab abnormalities, myocardial infarct, stroke, cancer, connective tissue diseases, etc.) including subjects with medical conditions that might require the use of immunosuppressive medications during the trial (e.g., severe asthma, rheumatoid arthritis, etc.).
* Subjects who have used exclusionary medications/treatments.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2004-08; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Evaluate degree of correction attainable with DL6049 compared to CosmoPlast Collagen Implant
in the treatment of dermal nasolabial fold wrinkles at 13 months following last application of study treatment.

SECONDARY OUTCOMES:
Treatment group comparisons at each timepoint of the treatment success rate (proportion of subjects with a photographic wrinkle severity grade of < 2), mean wrinkle severity grade, and investigator/subject global assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, MT, ASCP, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Brown SA, Rohrich RJ, Baumann L, Brandt FS, Fagien S, Glazer S, Kenkel JM, Lowe NJ, Monheit GD, Narins RS, Rendon MI, Werschler WP. Subject global evaluation and subject satisfaction using injectable poly-L-lactic acid versus human collagen for the correction of nasolabial fold wrinkles. Plast Reconstr Surg. 2011 Apr;127(4):1684-1692. doi: 10.1097/PRS.0b013e318208d371. PMID 21460676
- [Derived] Narins RS, Baumann L, Brandt FS, Fagien S, Glazer S, Lowe NJ, Monheit GD, Rendon MI, Rohrich RJ, Werschler WP. A randomized study of the efficacy and safety of injectable poly-L-lactic acid versus human-based collagen implant in the treatment of nasolabial fold wrinkles. J Am Acad Dermatol. 2010 Mar;62(3):448-62. doi: 10.1016/j.jaad.2009.07.040. PMID 20159311